CLINICAL TRIAL: NCT06436807
Title: Post-Market Clinical Follow-up Study to Assess the Safety, Performance, and Clinical Benefit of the CE-marked Drainova® ArgentiC Catheter
Brief Title: PMCF Study of the CE-marked Drainova® ArgentiC Catheter
Status: Recruiting | Type: Observational
Sponsor: ewimed GmbH (Industry)
Collaborators: LS medcap GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: 23-079
Record Dates: First submitted 2024-05-15; First posted 2024-05-31 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-07

CONDITIONS: Pleural Effusion; Pleural Effusion, Malignant; Ascites; Ascites, Malignant
MeSH Terms: conditions — Pleural Effusion; Pleural Effusion, Malignant; Ascites | interventions — Catheters, Indwelling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Device: Indwelling catheter — The tunneled catheter is an implant product that enables the drainage of effusion accumulations from serous body cavities so that the symptoms caused by an effusion are relieved by draining off the accumulated fluids.

SUMMARY:
The goal of this observational study is to learn about the performance of the drainova® ArgentiC Catheter in clinical routine, which is used to treat fluid accumulations in hollow body structures. The device is already on the market and participants receive the catheter as part of their regular treatment.

The main questions of this study are:

* Does the device function as intended?
* Are there any other safety risks that have not been identified?
* Does it lower the symptoms of the patients as intended?

Doctors and patients will answer questions regarding the improvement of the patients´ symptoms and if there were any problems with the catheter.

DETAILED DESCRIPTION:
The drainova® ArgentiC Catheter initially received the CE mark in 2019 under the Medical Device Directive 93/42/EEC, thus being considered a legacy device under the Medical Device Regulation (EU) 2017/745 (MDR). In order to fulfill the requirements of the MDR, this PMCF study is planned to be conducted to obtain clinical data on the device confirming its safety, performance and clinical benefit in clinical routine according to the instructions for use (IFU).

This PMCF study is performed as a purely observational activity within the current standards of care and without additional invasive or burdensome procedures. The drainova® ArgentiC catheter is a catheter indicated for the treatment of patients with pleural effusions and ascites, both in the malignant and non-malignant manifestations.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Patients being able to give informed consent

Exclusion Criteria:

Patients with any contraindication according to the IFU:

* presence of septa in the body cavity
* coagulopathy
* infection in the body cavity
* lymphatic effusion
* shift of the mediastinum (by more than 2 cm to the ipsilateral side of the pleural effusion)
* known allergies to any of the materials used in the drainage product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent, refractory, malignant and non-malignant effusions in serous body cavities according to the IFU.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Ascites- and pleural effusion-associated symptom relief | Discharge (1-7 days post-implantation)
  Measured by assessing the VAS score of the patient´s symptoms (e.g. pain) at baseline and discharge (defined by clinical routine).
Catheter patency | Discharge (1-7 days post-implantation)
  Occurrence of catheter blockage, occlusion or displacement
Implantation success | Immediately after procedure
  Must meet the following items:
  1. Successful placement at the defined location
  2. Feasibility of initial drainage of fluid (volume in ml)
Incidence of major adverse events, infections and device deficiencies | Up to three months post-implanatation
  Frequency of device- and/ or procedure-related major adverse events (MAEs), infections and device deficiencies

SECONDARY OUTCOMES:
Improvement of the patients´ quality-of-life vs. baseline | discharge (1-7 days post-implantation), 30 days, 3 months
  Quality-of-life will be assessed by QoL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Heidrun Steinle, Dr, Study Chair — LS medcap GmbH
Locations (11):
- Germany (11):
  - Universitätsklinikum Augsburg, Augsburg
  - Charité Universitätsmedizin Berlin, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Klinikum Chemnitz gGmbH MVZ Flemmingstraße, Chemnitz
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Clemenshospital, Münster
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Universitätsklinikum Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No